CLINICAL TRIAL: NCT05697159
Title: Exploiting Leading Edge 7 Tesla MRI Brain Imaging to Decipher Filgotinib's Mode of Analgesic Action in Rheumatoid Arthritis
Brief Title: 7 Tesla MRI Brain Imaging to Decipher Filgotinib's Mode of Analgesic Action in Rheumatoid Arthritis
Acronym: TEMPO
Status: Recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Other Study IDs: GN22RH315
Record Dates: First submitted 2022-12-15; First posted 2023-01-25 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis; Sickness Behavior; Inflammatory Disease; Autoimmune; Pain, Chronic
Keywords: Chronic pain; Rhuematoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Illness Behavior; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Research blood samples will be collected for peripheral immune phenotyping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an experimental medicine, single-centre, observational test-retest study to evaluate Filgotinib's mechanism of analgesic action in RA patients.

The investigators hypothesize that Filgotinib's mechanism of analgesic action is determined by at least two factors. The first is related to those CNS sensitization pathways seen in fibromyalgia, specifically DMN-insula brain functional connectivity and insular glutamate.

The second is related to peripheral inflammation, specifically joint synovitis, blood cytokines/chemokines and DAN-LIPL functional brain connectivity. The CNS sensitization pain pathways related to fibromyalgia are more quickly modified compared to those related to peripheral inflammation and help explain Filgotinib's rapid onset of effect.

DETAILED DESCRIPTION:
The revolution in rheumatoid arthritis (RA) therapeutics has been transformative for many patient outcomes. Yet most patients continue to experience life disabling pain. Strikingly, even those who achieve full disease remission with state-of-the-art anti-tumour necrosis factor (TNF) treatments report substantially higher levels of pain when compared to the general population. Such disconnect presents one of the greatest contemporary challenges to the care of patients with RA.

Considering the ongoing excess burden of pain in this patient population, trials of Janus kinase inhibitors (JAKinibs) present welcome data. JAKinibs deliver superior pain improvements in comparison to those receiving anti-TNF therapy. Of note, the majority of this effect has not been fully explained by markers of peripheral inflammation and remains to be understood. Moreover, JAKinibs appear to offer rapid analgesic benefit. Traditional DMARDS and modern biologics commonly take several weeks to bring relief whereas JAKinibs, such as filgotinib, begin to improve pain as early as 2 weeks, even before the observed attenuation of peripheral clinical inflammation.

In light of these clinical observations, the investigators believe that RA is a mixed pain state i.e., pain pathways exist in addition to established peripheral inflammatory nociceptive mechanisms. In particular, the central nervous system (CNS) may have an important role in determining RA pain. Recently our group were the first to delineate distinct neurobiological pain signatures in the brains of RA patients by employing functional connectivity magnetic resonance imaging (fcMRI) - a recent adaptation of functional MRI data that examines the synchrony of neural activity which modulates the efficiency and extent of neuronal transmission between brain regions. Specifically, the investigators identified and replicated two distinct pain signatures:

1. enhanced functional connectivity between the Default Mode Network (DMN) and insula, which was unrelated to levels of peripheral inflammation but, intriguingly, is an established neurobiological marker of fibromyalgia (the prototypical CNS pain sensitization disorder, and
2. enhanced functional connectivity between the Dorsal Attention Network (DAN) and the left inferior parietal lobule (LIPL) which was related to levels of peripheral inflammation.

Pre-clinical experiments have not only implicated the Janus kinase-signal transducer and activator of transcription (JAK-STAT) pathway with peripheral immune system functioning but also the brain. In the CNS, this pathway promotes gene expression associated with inflammation which in turn generates pro-nociceptive cytokines. However, there is now also emerging evidence to support the pathway's direct role in synaptic transmission and neurotransmitter receptor modulation. Specifically, the JAK-STAT pathway appears important in N-methyl-d-aspartate (NMDA) related synaptic plasticity - a ubiquitous glutamate receptor of the human brain. Their induction is selectively blocked by JAK inhibitors. Increases in glutamate and subsequent binding to NMDA receptors cause chaotic and incoherent neuronal functional activity. Human studies of fibromyalgia have consistently evidenced both elevated glutamate levels within the insula and dysfunctional neural connectivity. Moreover, fibromyalgia pharmacotherapy (pregablin), considered to reduce neural glutamate, rectifies both insular glutamate and brain functional connectivity (DMN-insula). JAK inhibition (JAKi) may facilitate the reduction of glutamate-NMDA binding and ultimately pain alleviation by normalising the functional activity of these same neural connections.

ELIGIBILITY:
Inclusion Criteria:

Patients with moderate to severe active RA who have been prescribed filgotinib in line with the Summary of Product Characterisation and are:

* Adults ≥18 years < 75 years.
* Right-handed (to reduce neuroimaging heterogeneity).

Exclusion Criteria:

* Inability to provide written informed consent.
* Severe physical impairment (e.g. blindness, deafness, paraplegia).
* Pregnant or breast feeding.
* Severe claustrophobia precluding MRI.
* Contraindications to MRI.
* Major confounding neurological disease including MS, Stroke, Traumatic Brain Injury.
* Previous targeted synthetic (e.g. baricitinib, tofacitinib) DMARD exposure for RA.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve 20 participants aged over 18 years with moderate to severe active RA, who have failed at least methotrexate, who fulfil the eligibility criteria below and who are scheduled to start Filgotinib as part of standard clinical practice. All will give full informed consent.
  The decision to commence filgotinib treatment, completion of all standard pre-biologic safety screening requirements, contraception requirements and patient consent to filgotinib treatment will be undertaken by the participant's usual care team as part of standard clinical practice and will be separate, and in advance of participation in this study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of Filgotinib in RA on CNS pain sensitisation (as measured by MRI brain) for DMN-Insula fMRI brain connectivity at 12 weeks. | 12 weeks
  Functional connectivity MRI (fMRI) investigations are conducted with subjects resting in the scanner. Ten minutes of whole-brain resting state fMRI data will be collected using a simultaneous-multi-slice (SMS) echoplanar-imaging (EPI) sequence of factor=3. A whole-brain T1-weighted structural image will also be collected using a twice magnetization-prepared rapid gradient echo (MP2RAGE) sequence. During the resting state, subjects will be instructed not to undertake any particular task and to stay awake with their eyes open on a fixation cross. Whole brain coverage will be performed.
  Upon collection of resting state fMRI data, pre-processing steps will include the removal of physiological artefacts, motion correction, realignment, registration, normalization and smoothing. Connectivity indices will be generated from matrices informed by our a priori determined regions of interest (DMN-Insula).
To evaluate the effects of Filgotinib in RA on CNS pain sensitisation (as measured by MRI brain) for insular glutamate levels at 12 weeks. | 12 weeks
  A magnetic resonance spectroscopy scan will be undertaken in order to detect the glutamate concentration. A single voxel sequence will be employed with semi-LASER preparation. A 20x20 mm3 voxel will be placed in the R posterior insula and shimming oA magnetic resonance spectroscopy scan will be undertaken in order to detect the glutamate concentration. A single voxel sequence will be employed with semi-LASER preparation. A 20x20 mm3 voxel will be placed in the R posterior insula and shimming of the static magnetic field will be performed using advanced methods best suited to MRS acquisition at 7T, such as FASTMAP. Spectra will be analysed and quantified in JMRUI or LCModel. In addition, multi-voxel techniques will be employed to provide quantitative maps of chemical concentration across the brain.

SECONDARY OUTCOMES:
To evaluate the effects of Filgotinib in RA on CNS pain sensitisation (as measured by MRI brain) for DMN-Insula fMRI brain connectivity at 4 weeks. | 0-4 weeks
  Functional connectivity MRI (fMRI) investigations are conducted with subjects resting in the scanner. Ten minutes of whole-brain resting state fMRI data will be collected using a simultaneous-multi-slice (SMS) echoplanar-imaging (EPI) sequence of factor=3. A whole-brain T1-weighted structural image will also be collected using a twice magnetization-prepared rapid gradient echo (MP2RAGE) sequence. During the resting state, subjects will be instructed not to undertake any particular task and to stay awake with their eyes open on a fixation cross. Whole brain coverage will be performed.
  Upon collection of resting state fMRI data, pre-processing steps will include the removal of physiological artefacts, motion correction, realignment, registration, normalization and smoothing. Connectivity indices will be generated from matrices informed by our a priori determined regions of interest (DMN-Insula).
To evaluate the effects of Filgotinib in RA on CNS pain sensitisation (as measured by MRI brain) for insular glutamate levels at 4 weeks. | 0-4 weeks
  A magnetic resonance spectroscopy scan will be undertaken in order to detect the glutamate concentration. A single voxel sequence will be employed with semi-LASER preparation. A 20x20 mm3 voxel will be placed in the R posterior insula and shimming oA magnetic resonance spectroscopy scan will be undertaken in order to detect the glutamate concentration. A single voxel sequence will be employed with semi-LASER preparation. A 20x20 mm3 voxel will be placed in the R posterior insula and shimming of the static magnetic field will be performed using advanced methods best suited to MRS acquisition at 7T, such as FASTMAP. Spectra will be analysed and quantified in JMRUI or LCModel. In addition, multi-voxel techniques will be employed to provide quantitative maps of chemical concentration across the brain.
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by MRI brain for DAN-LIPL fMRI brain connectivity (neurobiological marker of peripheral inflammatory pain) in the short term. | 0-4 weeks
  Functional connectivity MRI (fMRI) investigations are conducted with subjects resting in the scanner. Ten minutes of whole-brain resting state fMRI data will be collected using a simultaneous-multi-slice (SMS) echoplanar-imaging (EPI) sequence of factor=3. A whole-brain T1-weighted structural image will also be collected using a twice magnetization-prepared rapid gradient echo (MP2RAGE) sequence. During the resting state, subjects will be instructed not to undertake any particular task and to stay awake with their eyes open on a fixation cross. Whole brain coverage will be performed.
  Upon collection of resting state fMRI data, pre-processing steps will include the removal of physiological artefacts, motion correction, realignment, registration, normalization and smoothing. Connectivity indices will be generated from matrices informed by our a priori determined region of interest (DAN-IPL).
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by MRI brain for DAN-LIPL fMRI brain connectivity (neurobiological marker of peripheral inflammatory pain) in the medium term. | 12 weeks
  Functional connectivity MRI (fMRI) investigations are conducted with subjects resting in the scanner. Ten minutes of whole-brain resting state fMRI data will be collected using a simultaneous-multi-slice (SMS) echoplanar-imaging (EPI) sequence of factor=3. A whole-brain T1-weighted structural image will also be collected using a twice magnetization-prepared rapid gradient echo (MP2RAGE) sequence. During the resting state, subjects will be instructed not to undertake any particular task and to stay awake with their eyes open on a fixation cross. Whole brain coverage will be performed.
  Upon collection of resting state fMRI data, pre-processing steps will include the removal of physiological artefacts, motion correction, realignment, registration, normalization and smoothing. Connectivity indices will be generated from matrices informed by our a priori determined region of interest (DAN-IPL).
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by ultrasound joint, in the short term. | 0-4 weeks
  Rheumatoid arthritis is characterised by synovitis with symmetrical involvement. An ultrasound scan of pre-determined joints and up to 2 symptomatic joints with active disease will be performed at all visits. This will provide a robust surrogate measure of peripheral inflammation.
  The wrists, MCPs, PIPs joints of hands, knees, MTPs of both feet, and the 2 most symptomatic joints (if applicable) will be scanned and graded using the EULAR-OMERACT combined score. The ultrasonographic evaluation will further characterise the synovium involvement in the participants and will help to evaluate the response to treatment.
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by ultrasound joint, in the medium term. | 12 weeks
  Rheumatoid arthritis is characterised by synovitis with symmetrical involvement. An ultrasound scan of pre-determined joints and up to 2 symptomatic joints with active disease will be performed at all visits. This will provide a robust surrogate measure of peripheral inflammation.
  The wrists, MCPs, PIPs joints of hands, knees, MTPs of both feet, and the 2 most symptomatic joints (if applicable) will be scanned and graded using the EULAR-OMERACT combined score. The ultrasonographic evaluation will further characterise the synovium involvement in the participants and will help to evaluate the response to treatment.
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by blood cytokine/chemokines in the short term. | 0-4 weeks
  Research blood samples will be collected for peripheral immune phenotyping. This will consist of 10ml EDTA, 4ml EDTA, 8.5ml SST, and 2.5ml PAXgene RNA.
  An additional 5ml blood sample will be collected at each visit to allow calculation of the DAS28 score (CRP), unless this has been obtained by their standard care team within 14 days prior.
To evaluate the effects of Filgotinib in RA on peripheral inflammation related pain as measured by blood cytokine/chemokines in the medium term. | 0-12 weeks
  Research blood samples will be collected for peripheral immune phenotyping. This will consist of 10ml EDTA, 4ml EDTA, 8.5ml SST, and 2.5ml PAXgene RNA.
  An additional 5ml blood sample will be collected at each visit to allow calculation of the DAS28 score (CRP), unless this has been obtained by their standard care team within 14 days prior.
To evaluate the effects of Filgotinib in RA as measured by FACIT-F in the short term. | 0-4 weeks
  Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4)
  The FACIT-Fatigue Scale is a 13-item questionnaire to measure the level of participant fatigue from the past 7 days. Each item is scored on a scale from 0-4; (0 = very much fatigued, 4 = not at all fatigued).
To evaluate the effects of Filgotinib in RA as measured by FACIT-F in the medium term. | 0-12 weeks
  Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4)
  The FACIT-Fatigue Scale is a 13-item questionnaire to measure the level of participant fatigue from the past 7 days. Each item is scored on a scale from 0-4; (0 = very much fatigued, 4 = not at all fatigued).
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Anxiety in the short term. | 0-4 weeks
  Changes in anxiety as measured by the PROMIS-Anxiety
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Anxiety in the medium term. | 0-12 weeks
  Changes in anxiety as measured by the PROMIS-Anxiety
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Sleep related impairment in the short term. | 0-4 weeks
  Changes in sleep as measured by the PROMIS-Sleep related impairment.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Sleep related impairment in the medium term. | 0-12 weeks
  Changes in sleep as measured by the PROMIS-Sleep related impairment.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Pain interference in the short term. | 0-4 weeks
  Changes in pain interference as measured by the PROMIS-Pain inference.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Pain interference in the medium. | 0-12 weeks
  Changes in pain interference as measured by the PROMIS-Pain inference.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Fatigue in the short term. | 0-4 weeks
  Changes in fatigue as measured by the PROMIS-Fatigue.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Fatigue in the medium term. | 0-12 weeks
  Changes in fatigue as measured by the PROMIS-Fatigue.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Physical functioning short form in the short term. | 0-4 weeks
  Changes in physical functioning as measured by the PROMIS-Physical functioning short form from
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Physical functioning short form in the medium. | 0-12 weeks
  Changes in physical functioning as measured by the PROMIS-Physical functioning short form from
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Depression in the short term. | 0-4 weeks
  Changes in depression as measured by PROMIS-Depression.
To evaluate the effects of Filgotinib in RA on as measured by PROMIS-Depression in the medium term. | 0-12 weeks
  Changes in depression as measured by PROMIS-Depression.
To evaluate the effects of Filgotinib in RA as measured by the McGill Pain Questionnaire in the short term. | 0-4 weeks
  A Short-Form McGill Pain Questionnaire consisting of three sections.
  The first part consists of 15 items that describe qualities of pain. Participants score each item within a range of 0-3 (0 = none, 1 = mild, 2 = moderate, 3 = severe) based on their experience from the past seven days.
  The second part contains a 100 mm visual analogue scale where participants place a vertical line in the position that best describes their pain during the past seven days, from 'No Pain' to 'Worst Possible Pain'.
  The third part measures present pain intensity on a scale of 0-5 (0 = No Pain, 1 = Mild, 2 = Discomforting, 3 = Distressing, 4 = Horrible, 5 = Excruciating).
To evaluate the effects of Filgotinib in RA as measured by the McGill Pain Questionnaire in the medium term. | 0-12 weeks
  A Short-Form McGill Pain Questionnaire consisting of three sections.
  The first part consists of 15 items that describe qualities of pain. Participants score each item within a range of 0-3 (0 = none, 1 = mild, 2 = moderate, 3 = severe) based on their experience from the past seven days.
  The second part contains a 100 mm visual analogue scale where participants place a vertical line in the position that best describes their pain during the past seven days, from 'No Pain' to 'Worst Possible Pain'.
  The third part measures present pain intensity on a scale of 0-5 (0 = No Pain, 1 = Mild, 2 = Discomforting, 3 = Distressing, 4 = Horrible, 5 = Excruciating).
To evaluate the effects of Filgotinib in RA on as measured by Global Impression of Change in the short term. | 0-4 weeks
  Participant selects an option to describe their impression of change with regards to their RA since entering the study.
  Options are: Very Much Improved, Much Improved, Slightly Improved, No Change, Much Worse, Very Much Worse.
To evaluate the effects of Filgotinib in RA on as measured by Global Impression of Change in the medium term. | 0-12 weeks
  Participant selects an option to describe their impression of change with regards to their RA since entering the study.
  Options are: Very Much Improved, Much Improved, Slightly Improved, No Change, Much Worse, Very Much Worse.
To evaluate the effects of Filgotinib in RA as measured by Cognitive Failures Questionnaire in the short term. | 0-4 weeks
  Cognitive Failures Questionnaire consists of 25 items corresponding to changes in cognitive functions, with a range of 4-0 (4 = Very Often; 3 = Quite Often; 2 = Occasionally; 1 = Very rarely; 0 = Never) to determine their frequency.
To evaluate the effects of Filgotinib in RA as measured by Cognitive Failures Questionnaire in the medium term. | 0-12 weeks
  Cognitive Failures Questionnaire consists of 25 items corresponding to changes in cognitive functions, with a range of 4-0 (4 = Very Often; 3 = Quite Often; 2 = Occasionally; 1 = Very rarely; 0 = Never) to determine their frequency.
To evaluate the effects of Filgotinib in RA on as measured by the Sickness Questionnaire in the short term. | 0-4 weeks
  The sickness questionnaire is a 10-item instrument used to capture perceived sickness behaviour. It was developed to display sensitivity to an inflammatory challenge and have adequate psychometric properties.
To evaluate the effects of Filgotinib in RA on as measured by the Sickness Questionnaire in the medium term. | 0-12 weeks
  The sickness questionnaire is a 10-item instrument used to capture perceived sickness behaviour. It was developed to display sensitivity to an inflammatory challenge and have adequate psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Basu, MD, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Neil Basu, Glasgow, United Kingdom

REFERENCES:
- [Background] Basu N, Kaplan CM, Ichesco E, Larkin T, Harris RE, Murray A, Waiter G, Clauw DJ. Neurobiologic Features of Fibromyalgia Are Also Present Among Rheumatoid Arthritis Patients. Arthritis Rheumatol. 2018 Jul;70(7):1000-1007. doi: 10.1002/art.40451. Epub 2018 May 11. PMID 29439291
- [Background] D'Agostino MA, Terslev L, Aegerter P, Backhaus M, Balint P, Bruyn GA, Filippucci E, Grassi W, Iagnocco A, Jousse-Joulin S, Kane D, Naredo E, Schmidt W, Szkudlarek M, Conaghan PG, Wakefield RJ. Scoring ultrasound synovitis in rheumatoid arthritis: a EULAR-OMERACT ultrasound taskforce-Part 1: definition and development of a standardised, consensus-based scoring system. RMD Open. 2017 Jul 11;3(1):e000428. doi: 10.1136/rmdopen-2016-000428. eCollection 2017. PMID 28948983
- [Background] Schrepf A, Kaplan CM, Ichesco E, Larkin T, Harte SE, Harris RE, Murray AD, Waiter GD, Clauw DJ, Basu N. A multi-modal MRI study of the central response to inflammation in rheumatoid arthritis. Nat Commun. 2018 Jun 8;9(1):2243. doi: 10.1038/s41467-018-04648-0. PMID 29884867